CLINICAL TRIAL: NCT00440271
Title: SPRING: Safety, Efficacy, Pharmacokinetics of tipRanavi/r IN Race/Gender HIV+ Patients Randomized to Therapeutic Drug Monitoring or Standard of Care
Brief Title: SPRING: Safety, Efficacy, Pharmacokinetics of tipRanavir/r IN Race/Gender HIV+ Patients Randomized to TDM or SoC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.98; EudraCT No.: 2005-005264-86
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Enfuvirtide; Maraviroc; Raltegravir Potassium

ARMS (2):
- Standard of Care (SoC) (Other): Standard of Care (SOC) Arm = Tipranavir/ritonavir (TPV/r) capsules taken orally at a dose of 500 mg/200 mg twice a day (BID) plus optimized background regimen (OBR). No TPV/r dose changes were permitted.
  Interventions: Drug: tipranavir; Drug: ritonavir; Drug: Optimized Background Regimen (OBR)
- Therapeutic Drug Monitoring (TDM) (Other): Therapeutic Drug Monitoring (TDM) Arm = Patients began by receiving standard of care (SOC) tipranavir/ritonavir (TPV/r) capsules orally at a dose of 500 mg/200 mg twice a day (BID) plus optimized background regimen (OBR) followed, if needed, by TPV or ritonavir (RTV) dose adjustments at Week 4, 6, 10, 14, 18, 22, 26 and 30 based on viral response, phenotypic inhibitory quotient (IQ), and TPV trough concentrations.
  Interventions: Drug: tipranavir; Drug: ritonavir; Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Drug: tipranavir
Drug: ritonavir
Drug: Optimized Background Regimen (OBR) — Patients received between two and four active anti-retroviral medications based on resistance testing results, as background treatment, and remained on these for the duration of the trial.
  Other Names: Nucleoside Reverse Transcriptase Inhibitors (NRTIs),; Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs),; Enfuvirtide,; Maraviroc,; Raltegravir

SUMMARY:
The primary purpose of this study is to:

1. Demonstrate the safety and efficacy of tipranavir/ritonavir (TPV/r) among a racially diverse HIV+ population (males and females) who are three-class (nucleoside reverse transcriptase inhibitor (NRTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), and protease inhibitor (PI)) experienced with documented resistance to more than one PI.
2. Determine pharmacokinetic data in this racially and gender diverse population.
3. Determine the potential utility of using therapeutic drug monitoring (TDM) in improving efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria for the study are:

1. HIV-1 infected adults, men and women at least 18 years of age.
2. 3-class (nucleoside reverse transcriptase inhibitor (NRTI), non-nucleoside reverse transcriptase inhibitor (NNRTI), and protease inhibitor (PI)) treatment-experienced (min of 3-months duration for each class) with resistance to more than one PI (on screening resistance testing). NNRTI-naïve patients who have genotypically documented NNRTI-resistance mutations on past or screening resistance testing would be eligible.
3. CD4+ T lymphocyte count >=50 cells/mm3.
4. HIV-1 viral load >=1,000 copies/mL at screening.
5. The antiretroviral (ARV) study treatment regimen must consist of TPV/r in combo with an optimized background regimen (OBR) of 2-4 agents: N(t)RTIs (NRTI or NtRTI), enfuvirtide (ENF), and/or, where available, a trial approved expanded access program (EAP) investigational agent.
6. Acceptable screening laboratory values that indicate adequate baseline organ function.
7. Acceptable medical history with a chest X-ray without evidence of active disease and an electrocardiogram (ECG) without clinically important abnormalities within one year of the study.
8. A reliable method of barrier contraception will be used by all female patients who are of childbearing potential.

Exclusion Criteria:

Main exclusion criteria for the study are:

1. Known hypersensitivity to the tipranavir (TPV) or ritonavir (RTV).
2. ARV medication naïve.
3. Genotypic resistance to TPV (defined as a TPV mutation score >7).
4. Patients on recent drug holiday, defined as off antiretroviral (ARV) medications for at least 7 consecutive days within the month prior to screening.
5. Prior tipranavir use.
6. Inability to adhere to the requirements of the protocol.
7. Patients with prior history of hemorrhagic stroke or intracranial aneurysm.
8. Patients with a history of ischemic stroke, neurosurgery or skull trauma within 4 weeks prior to screening.
9. History of Progressive Multifocal Leukoencephalopathy, Visceral Kaposi's Sarcoma, and/or any malignancy.
10. Any acquired immunodeficiency syndrome (AIDS) defining illness that is unresolved, symptomatic or not stable on treatment for at least 12 weeks at screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- United States (16):
  - 1182.98.033 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.98.018 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1182.98.014 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1182.98.041 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1182.98.004 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1182.98.002 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1182.98.016 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.98.026 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.98.034 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1182.98.040 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1182.98.006 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1182.98.007 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1182.98.020 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1182.98.029 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1182.98.023 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1182.98.009 Boehringer Ingelheim Investigational Site, Houston, Texas
- Argentina (3):
  - 1182.98.5405 CENTRO de INFECTOLOGIA y ASISTENCIA (CIAS), Capital Federal ,Buenos Aires
  - 1182.98.5403 Centro Hospital Higa - Dr Oscar Alende, Mar del Plata
  - 1182.98.5402 Caici, Rosario
- Brazil (4):
  - 1182.98.55002 Hospital DIA, Sacomã - São Paulo
  - 1182.98.55004 Unidade de Referência em doenças Infecciosas Preveníveis, Santo André
  - 1182.98.55001 Universidade Federal de Sao Paulo, São Paulo
  - 1182.98.55003 Centro de Referência e Treinamento - DST/AIDS, Vila Mariana - Sao Paulo
- 1182.98.1007 Boehringer Ingelheim Investigational Site, Quebec, Ste Foy, Quebec, Canada
- Germany (2):
  - 1182.98.4903 Boehringer Ingelheim Investigational Site, Bochum
  - 1182.98.4908 Boehringer Ingelheim Investigational Site, Hamburg
- 1182.98.3907 Boehringer Ingelheim Investigational Site, Torino, Italy
- Spain (3):
  - 1182.98.3402, Barcelona
  - 1182.98.3405, Madrid
  - 1182.98.3406, Madrid

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Started | 15 | 18
Completed | 3 | 3
Not Completed | 12 | 15
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Due to closure of trial | 8 | 10
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM) | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (8.2) | 43.2 (10.6) | 44.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response at Week 48
Description: percentage of participants whose viral load <50 copies/mL at Week 48
Time Frame: after 48 weeks of treatment
Population: The study was terminated early due to low patient enrollment, and, therefore, no analysis was performed on the primary and secondary endpoints.
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants Whose Viral Load <50 Copies/mL at Each Visit Including Visits at Weeks 24 and 48
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants Whose Viral Load <400 Copies/mL at Each Visit Including Visits at Weeks 24 and 48
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Whose ≥1 log10 Drop in Viral Load From Baseline at All Visits, Including Visits at Weeks 24 and 48
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Viral Load From Baseline at Each Visit
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Treatment Failure
Description: For patients who never achieve a confirmed virologic response, time to treatment failure is defined as 0. For patients who achieve a confirmed virologic response, time to treatment failure is the earliest time of either: death, permanent discontinuation of the study drug or loss to follow-up, introduction of a new anti-retroviral drug to the regimen if it is not solely related to either toxicity or intolerance clearly attributable to a background drug, but not the study drug, or first occurrence of a VL >50 copies/mL at two consecutive measurements after having achieved a VL <50 copies/mL.
Time Frame: after Day 1 of treatment
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to New AIDS or AIDS Related Progression Event or Death
Time Frame: after Day 1 of treatment
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in CD4+ and CD8+ Cell Counts From Baseline at Each Visit Including Visits at Week 24 and Week 48
Time Frame: after 2 weeks of treatment till Week 48 (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Ratio of CD38+/CD8+ From Baseline to Week 48
Time Frame: after 2 weeks of treatment till Week 48 (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Tipranavir (TPV) and Ritonavir (RTV) Trough Concentrations at Week 2, Week 4, Week 8, Week 12, Week 24, Week 36 and Week 48
Time Frame: after 2 weeks of treatment till Week 48 (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Patients Adherence With Study Medication Based on Pill Count
Time Frame: after 4 weeks of treatment
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Occurrence of TPV Inhibitory Quotient (IQ) >60 at Each Visit Where TPV Concentration is Measured
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Occurrence of TPV Trough Concentration >120 μM
Time Frame: after 2 weeks of treatment (Weeks 2, 4, 8, 12, 24, 36, and 48)
Population: as for outcome 1
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Post-dose TPV and RTV Concentrations at Week 4
Time Frame: Week 4
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 weeks of treatment plus 30 days follow-up
Description: MedDra 11.1 WHO-DD 08SEP
Arm/Group | Standard of Care (SoC) | Therapeutic Drug Monitoring (TDM)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 12/15 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (SoC) (N=15) | Therapeutic Drug Monitoring (TDM) (N=18)
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Adverse drug reaction (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Feeling abnormal (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 1
Blood amylase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to low patient enrollment, and, therefore, no analysis was performed on the primary and secondary endpoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract